CLINICAL TRIAL: NCT05995899
Title: An Open-label, Single Center Investigator Sponsored Study Assessing the Effect of Tenapanor on Metagenomic and Metabolomic Markers in Patients With Irritable Bowel Syndrome With Constipation
Brief Title: Effect of Tenapanor on the Metagenomics and Metabolomics of Patients With Irritable Bowel Syndrome With Constipation
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Kyle Staller, MD, MPH (Other)
Collaborators: Ardelyx (Industry)
Responsible Party: Sponsor-Investigator, Kyle Staller, MD, MPH, Gastroenterology Physician, Massachusetts General Hospital
Organization: Massachusetts General Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023P001911
Record Dates: First submitted 2023-08-03; First posted 2023-08-16 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-09

CONDITIONS: IBS; IBS - Irritable Bowel Syndrome
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — tenapanor

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Patients with IBS-C (Experimental)
  Interventions: Drug: Tenapanor

INTERVENTIONS:
Drug: Tenapanor — IBS-C patients will ingest one capsule of tenapanor (50 mg per dose), twice daily, before breakfast and dinner for a total of 8 weeks

SUMMARY:
The aim of this study is to better understand how tenapanor affects the metagenomics and metabolomics of patients with irritable bowel syndrome with constipation (IBS-C). Tenapanor is the newest FDA-approved agent for IBS-C. It is a small molecule that inhibits the NHE3 receptor, leading to impaired sodium and water absorption in the intestine. Previous clinical trials comparing tenapanor to placebo showed that a 50 mg dose of tenapanor led to increased bowel movements and decreased abdominal pain. This study consists of an 8-week treatment period in which subjects will ingest one capsule of tenapanor (50 mg per dose), twice daily, and send in stool samples following 4 weeks and 8 weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Ages 18-75 years old
2. BMI >18.5 and <35 kg/m2
3. Rome IV criteria for IBS-C for at least 6 months
4. Compliant with baseline stool submission prior to initiation of medication
5. Ability to follow verbal and written instructions
6. Ability to record daily bowel habits, including frequency, stool consistency (BSFS), and symptom severity
7. Willingness to avoid major dietary changes and use of probiotics during the study period
8. Informed consent form signed by the subjects

Exclusion Criteria:

1. History of loose stools
2. History of irritable bowel syndrome with diarrhea (IBS-D) or mixed irritable bowel syndrome (IBS-M)
3. Non-compliance with baseline stool submission
4. Previous use of tenapanor
5. GI motility obstruction or GI tract structural abnormality
6. Current use of prescribed or illicit opioids
7. History of pelvic floor dysfunction
8. Need for manual maneuvers in order to achieve a BM
9. History of GI lumen surgery at any time or other GI or abdominal operations within 60 days prior to entry into the study
10. History of high-dose stimulative or cathartic laxative abuse as judged by investigator team
11. Severe IBS-C as judged by the investigator
12. Neurological disorders, metabolic disorders, or other significant disease that would impair their ability to participate in the study
13. Cardiovascular disease, diabetes, cancer, Crohn's disease, ulcerative colitis
14. BMI of <18.5 or >35 kg/m2
15. Pregnancy (or positive serum or urine pregnancy test(s) in females of childbearing potential) or lactation
16. Absence of contraception in females of childbearing potential
17. History of allergic reaction to tenapanor
18. Administration of other FDA-approved agents for the treatment of IBS-C within 1 month prior to Screening Visit:

    * Linaclotide
    * Lubiprostone
    * Plecanatide
19. If treated with any of the following medications, dosing (or approximate frequency of 'as needed' use) must be stable for at least 30 days prior to Screening Visit and the subject must agree to maintain the same dose (or approximate frequency of 'as needed' use) or a decreased dose of medication throughout the study:

    * Probiotics
    * Bulk laxatives, fiber, and stool softeners
20. Exclusion of colonic inertia with symptoms of < 1 BM per 2 weeks
21. Subjects anticipating surgical intervention during the study
22. Known history of diabetes (type 1 or 2)
23. Subjects with recent antibiotic use (last 3 months) or anticipated antibiotic use during the study period
24. History of inflammatory bowel disease
25. Supine SBP > 160 mm Hg and/or supine DBP > 95 mm Hg (mean of two consecutive readings)
26. Angina, coronary bypass, or myocardial infarction within 6 months prior to Screening Visit
27. History of swallowing disorders
28. History of gastric bypass or any other gastric surgery
29. History of small bowel resection (except if related to appendectomy)
30. History of gastric or duodenal ulcer
31. History of gastroparesis
32. History of abdominal radiation treatment
33. History of pancreatitis
34. History of intestinal stricture (e.g., Crohn's disease)
35. History of intestinal obstruction or subjects at high risk of intestinal obstruction including suspected small bowel adhesions
36. History of malabsorption
37. History of hepatitis B or C
38. History of human immunodeficiency virus
39. History of cancer within the past 5 years (except adequately-treated localized basal cell skin cancer or in situ uterine cervical cancer)
40. Any other clinically significant disease interfering with the assessments of tenapanor, according to the Investigator (e.g., disease requiring corrective treatment, potentially leading to study discontinuation)
41. HbA1c > 8.5% (> 69 mmol/mol)

43. Any relevant biochemical abnormality interfering with the assessments of tenapanor, according to the Investigator 44. Antidiabetic medications within 1 month prior to Screening Visit (except stable dose of metformin, ≤ 1500 mg/day, for at least 1 month in subjects with type 2 diabetes) 45. Medications requiring mandatory administration twice per day with meals

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-02-06 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Measuring metagenomics of stool samples using whole genome shotgun sequencing (WGS) | Subjects will submit stool samples at 0 weeks, 4 weeks, and 8 weeks following treatment.
  Sequence-based microbial community surveys will be carried out by whole genome shotgun sequencing (WGS) at the Broad Institute using their established sequencing and analysis pipeline for the Illumina HiSeq2000 platform used in Human Microbiome Project (HMP) to characterize rare taxa and understand relationships between community membership and function. Composition analysis of metagenome will be performed using the read-based bioinformatics analysis suite. Functional genomic profiles, detailed species-specific reconstruction of microbial metabolic pathways, their complement of gene orthologs, taxonomic distributions, and abundances will be generated with HUMAnN2. This will provide taxon-specific profiles of UniRef orthologous gene families, MetCyc, UniPathway, and KEGG pathways to survey microbial community metabolite production potential in each metagenome according to tenapanor use.
Measuring metabolomics of stool samples using the DiscoveryHD4TM Platform | Subjects will submit stool samples at 0 weeks, 4 weeks, and 8 weeks following treatment.
  Stool samples will also undergo metabolomics profiling at Metabolon Inc using the DiscoveryHD4TM Platform, a comprehensive and well-validated high-throughput metabolomics platform available for clinical and research use. Metabolites are identified by automated comparison of the ion features in the experimental samples to a reference library of ~8,000 chemical standard entries that include retention time, molecular weight (m/z), preferred adducts, in-source fragments and MS spectra, and they are visually curated for quality control using Metabolon software.

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States